CLINICAL TRIAL: NCT02175875
Title: The Effect of Antithrombotic Treatment Administrated Through Nasogastric Tubes to Comatose Patients Undergoing Acute Percutaneous Coronary Intervention
Brief Title: Ticagrelor for the Comatose
Acronym: TICOMA
Status: Completed | Type: Observational
Sponsor: Lene Holmvang (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Lene Holmvang, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: EudraCT nr: 2013-005529-22; 2013-005529-22 (EudraCT Number)
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Comatose
Keywords: ticagrelor; platelet function test; comatose; PCI; naso-gastric tube
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- comatose patients: 180 mg ticagrelor followed by 90 mg BID for comatose patients after cardiac arrest

SUMMARY:
The study will investigate the effect of the oral antiplatelet agent ticagrelor (Brilique) when it is administrated through a nasogastric tube in comatose patients. The platelet function can be determined by various platelet function tests (PFT), Multiplate and VerifyNow . As control, the reference intervals from the literature are used. Futhermore, plasma concentrations of the active metabolite will be determined at aeveral timepoints after first intake of a bolus dose.

DETAILED DESCRIPTION:
Study population:

Fifty patients admitted after cardiac arrest and who have all undergone acutte PCI will be inclded in the trial.

All patients hospitalized at the cardiologic intensive department, RH, who are receiving ticagrelor (Brilique) through a nasogastric tube can be enrolled in the study. Administration of ticagrelor will follow usual indications and will thus only be used for patients considered to suffer from acute coronary syndromes (ACS). Blood samples are collected from an already inserted central venous catheter (CVC) and will therefore not affect the patients any further. The first samples will be collected directly before the first doses of medicine is given (t0), the samples are thereafter being repeatedly taken after (2(±1), 4(±1), 8(±1),12(±1), and 24(±2) hours, hereafter daily (kl. 6-8 am) until after the first day where the patient can receive tablets orally, or until intensive care treatment is terminated (though, at most 5 days of sampling, addition to the first day).

Medical treatment

All study participants will be receiving antithrombotic treatment on clinical indication: aspirin + ticagrelor (brilique), thus no antithrombotic is given without indication and doses (bolus and maintain dose) is given according to the product information. Time sets for medicine administration is controlled by the EPM (electronic patient medication module). The Ticagrelor used is "medicine-off-the-shelf" administrated in following doses:

Ticagrelor: bolus 180 mg p.o. as soon as possible after PCI and after insertion of a naso-gastic tube. Maintenance doses (90 mg) are administrated at 6 AM (+/- 1h) and 6PM (+/- 1h) with the first maintenance dose administrated < 12 hours after bolus a 6AM or 6 PM whatever comes first. Contraindications as stated in the respectively product's summary are followed.

Blood samples Blood collected for platelet function analysis are analysed immediately by VerifyNow and Multiplate and TEG-platelet mapping if available. In addition, 50 ml of blood is saved in a research bio bank for a collected analysis of concentrations of ticagrelor (active metabolite and parent compound) at the end of study. Residual blood will be destroyed. The maximum total amount of blood collected will be 150 ml.

Informed consent in a trial of in-capacitated patients In the trial, patients who all are unconscious due to prior cardiac arrest or due to cardiogenic shock are participating. Most of the patients will be connected to life support and others are in unconscious states, which exclude the possibility of obtaining an informed agreement. All patients are > 18 years old.

The study will be conducted under Danish and international guidelines for good clinical practice (ICHP-GCP) and the study are approved by the regional scientific ethical committee and the Danish Medical Agency. The participating study persons will all be unconscious, sedated or in a cerebral situation where you cannot reasonable consider involvement in a scientific study, and they are therefore not able to give informed consent in the acute phase. Current guidelines recommend acute revascularization and if necessary, circulation support and/or a cooling regimen and all treatment will be in accordance with local practice Inclusion in the project before obtaining informed consent can be justified according to the committee law's § 12. There are established a committee of two "legal guardians" (Danish: forsøgsværge), who have to agree to the patient's involvement in the trial and will make an individual judgement of the single patient's suitability to participate. The "legal guardian" (Danish: forsøgsværge) will at the time, receive the updated study protocol and all the information material which otherwise would have been presented to the patient/next of kin in the context of obtaining informed consent.

Study procedures can start after accept from the legal guardian (Danish:forsøgsværge) however subsequent informed consent from the patient's next-of-kin should be obtained as soon as possible, as well as from the patient's general practitioner/health officer.

Patients who regain their conscious will be asked for informed agreement. The agreeing part will be provided with information in word and speech regarding the study, so as the concerned will be able to make an informed decision about participation in the trial. The concerned part will be informed by the, for the study responsible, doctor or the attending doctor, who will be trained in the protocol. The declaration of consent has to be signed by the patient himself or his/her next-of-kin, as well as by the investigator who obtains the informed agreement.

ELIGIBILITY:
Inclusion criteria are for the trial are:

1. Recent (<3 hours) PCI and therefore indication for oral ADP inhibitor treatment
2. The patient is in a condition that disables normal oral administration of tablets and requires naso-gastric tube insertion.

Exclusion criteria

1. Age < 18 years old
2. Serious bleeding tendency, absolute contraindication to antithrombotic treatment (as defined in product information)
3. Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 50 unconscious patients, primary due to cardiac arrest or cardiogenic shock. All patients have been undergoing recent percutaneous coronary intervention (PCI) and are hospitalized at the cardiac intensive care unit.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Platelet inhibition measured by VerifyNow at 12 hours | 12 hours after ticagrelor bolus

SECONDARY OUTCOMES:
Platelet inhibition at several time points by VerifyNow and Multiplate | 2hours to 5 days after admission

OTHER OUTCOMES:
Plasma concentration of active drug and parent compound | 2 hours to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Lene Holmvang, MD, PHD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen O, Denmark